CLINICAL TRIAL: NCT03836859
Title: Phase I, Randomized, Double-masked, Placebo-controlled Study (6 Days) to Evaluate the Safety, Tolerability and Pharmacokinetics of Recombinant Human Nerve Growth Factor Eye Drops in Healthy Male and Female Volunteers of Japanese Ethnicity
Brief Title: Study to Evaluate Safety, Tolerability & PK of rhNGF in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0117
Record Dates: First submitted 2018-07-19; First posted 2019-02-11 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: Tolerability and PK
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (subject, Investigator, site staff and Sponsor's clinical research personnel)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhNGF 20μg/mL (Experimental): rhNGF 20μg/mL eye drop solution, formulation containing L-methionine as excipient.
  Interventions: Drug: rhNGF 20μg/mL
- Placebo (Placebo Comparator): Vehicle: formulation containing L-methionine as excipient.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: rhNGF 20μg/mL — Study Eye (For subjects randomized to rhNGF group) Day 1: One drop instilled into study eye (35 μL, corresponding to 0.70 μg of rhNGF).
  Day 2, 3, 4, 5, 6: One drop six times a day (every 2h) into study eye (210 μL, corresponding to 4.20 μg of rhNGF).
  Total dose in the study eye will be 31 drops (1085 μL, equivalent to 21.7 μg rhNGF) over 6 days.
  Other Names: cenegermin
  Arms: rhNGF 20μg/mL
Other: Placebo — Vehicle: formulation containing L-methionine as excipient.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of a single short-term and a multiple dose scheme of rhNGF when administered as eye drops in healthy subjects of Japanese ethnicity.

The secondary objective of this study is to assess the pharmacokinetics of single and multiple doses of rhNGF when administered as eye drops in healthy subjects of Japanese ethnicity.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-masked, placebo-controlled eye drops administration study of rhNGF in healthy male and female subjects of Japanese Ethnicity to evaluate the Safety, Tolerability and Pharmacokinetics of Recombinant Human Nerve Growth Factor Eye Drops (rhNGF 20 μg/mL -formulation containing L-methionine as excipient) versus vehicle (vehicle control containing L-methionine as excipient) in Healthy Male and Female Volunteers of Japanese Ethnicity. The IMP was administered in the study Eye with the following scheme:

Day 1: One drop instilled into study eye (35 μL, corresponding to 0.70 μg of rhNGF).

Day 2, 3, 4, 5, 6: One drop six times a day (every 2h) into study eye (210 μL, corresponding to 4.20 μg of rhNGF).

Total dose in the study eye will be 31 drops (1085 μL, equivalent to 21.7 μg rhNGF) over 6 days.

The reference product (vehicle) was administered in the study eye with the following scheme:

Day 1: One drop instilled into study eye (35 μL, corresponding to 0 μg of rhNGF].

Day 2, 3, 4, 5, 6: One drop six times a day (every 2h) into study eye (210 μL, corresponding to 0 μg of rhNGF).

A total dose of placebo vehicle in the study eye will be 31 drops (1085 μL, 0 μg rhNGF) over 6 days.

For the Fellow (Non-Study) Eye for all subjects, the scheme was the following:

Day 1: One drop instilled into a fellow eye (35 μL, corresponding to 0 μg of rhNGF).

Day 2, 3, 4, 5, 6: One drop six times a day (every 2h) into a fellow eye (210 μL, corresponding to 0 μg of rhNGF).

A total dose of placebo vehicle in the fellow eye will be 31 drops (1085 μL, 0 μg rhNGF) over 6 days.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each subject must fulfil the following inclusion criteria.Each subject must meet all of the following inclusion criteria at the pre-study Screening visit (within 20 days prior to admission in the Unit for the dosing period) in order to participate in this study.

1. Male or female subjects of Japanese ethnicity, aged between 18 and 60 years inclusive, who must have all four Japanese grandparents who were born in Japan.
2. Subject has to be able to communicate well with the investigator, understands and complies with the requirements of the study, and understands and signs the written volunteer informed consent form.
3. Subject's systemic and ocular medical history must be considered normal in the opinion of the investigator at the Screening and Baseline visits.
4. Subject with Best corrected distance visual acuity (BCDVA) score ≥83 ETDRS letters, ≤ 0.00 LogMAR [20/20 Snellen or 1.0 decimal fraction] in each eye at the Screening and Baseline visits.
5. Normal anterior segment on external and slit lamp examination in both eyes at the Screening and Baseline visits.
6. Normal posterior segment on fundus ophthalmoscopic examination in both eyes at the Screening and Baseline visits.
7. Subject must be considered in good systemic health in the opinion of the investigator at the Screening and Baseline visits, as determined by:

   1. Subject's body mass index is between 18.5 and 30.4 kg/m2 inclusive
   2. A pre-study physical examination with no clinically significant abnormalities.
   3. Vital signs within clinically acceptable ranges for the purposes of the study (sitting systolic blood pressure [BP] ≥ 90 mmHg and ≤ 150 mmHg; diastolic BP ≥ 50 mmHg and ≤ 95 mmHg; heart rate ≥ 40 and ≤ 100 beats per minute; oral body temperature ≥ 35.5°C and ≤ 37.5°C).
   4. An ECG with no clinically significant abnormalities.
   5. Pre-study clinical laboratory findings within normal range or not deemed clinically significant in the opinion of the investigator if outside of the normal range
8. Woman subject who meets the criteria for post-menopausal stage (post menopause is defined as the period following peri-menopause, i.e. postmenopausal after 12 months without a menstrual period and with a serum FSH value within the reference range for postmenopausal females at Screening) or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy) or woman subject using oral, injected or implanted hormonal methods of contraception or with a double barrier methods of contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. A female condom and a male condom should not be used together as friction between the two can result in either product failing.
9. Male subjects with female partners of child-bearing potential must use 2 different forms of highly effective contraception throughout the study and for a further 3 months after the follow-up visit and all male subjects must be willing to avoid donating sperm during this time. The following methods of contraception are considered to be highly effective: established use of oral, injected or implanted hormonal contraception; placement of an intrauterine device or intrauterine system; use of a barrier method of contraception (condom or occlusive cap with use of a spermicide); male sterilisation (post-vasectomy documentation of the absence of sperm in the ejaculate must be provided).

Exclusion Criteria:

Subjects meeting any of the following criteria at Screening will be excluded from entry into the study:

1. Subject has had a clinically significant illness in the 6 weeks before screening in the opinion of the investigator.
2. Subject is not suitable to participate in the study in the opinion of the investigator
3. Subject has participated in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
4. Subject has had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or has a clinically significant allergy to drugs, foods or other materials (in the opinion of the investigator).
5. Administration of any topical ocular (prescription or over the counter including artificial tears) or systemic medication including herbal product or fish oil preparations within 14 days before the first dose of study drug. Vitamins and mineral supplements not containing other substances are allowed until 96 hours before each dose if considered by the Investigator unlikely to interfere with the study results. Paracetamol at doses of at most 2 grams per day and ibuprofen at doses of at most 1200 mg per day for no more than 3 consecutive days or 6 non-consecutive days are allowed. Oral, injectable and implantable hormonal contraceptives are allowed without restrictions for female subjects. Longer exclusion periods apply for:

   1. amiodarone and hydroxychloroquine (210 days),
   2. monoclonal antibodies/ immunoglobulins/ other therapeutic proteins (120 days)
   3. Experimental drugs with a half life known to the Study Unit: Five half lives plus 2 weeks
   4. Experimental drugs with a half-life unknown to the Study Unit: 120 days
   5. chloroquine and flunarizine (100 days)
   6. fluoxetine (75 days),
   7. benzodiazepines different from midazolam, lorazepam and triazolam, chlorpromazine, mephenytoin, nortryptyline, phenobarbital, primidone, carbamazepine, phenytoin and phenprocoumon (35 days).
6. Subject has a significant history of drug/solvent abuse or a positive drugs of abuse test at any time during the study.
7. Subject has a history of alcohol abuse or currently drinks in excess of 28 units per week or has a positive alcohol breath test at any time during the study.
8. Subject is a smoker or has smoked in the 6 months prior to dosing.
9. Subject who has a positive human immunodeficiency virus (HIV) screen, hepatitis B screen or hepatitis C screen.
10. Subject has donated blood or blood products (e.g., plasma or platelets) within the 3 months prior to screening.
11. Subject has a partner who will be pregnant or breastfeeding during the study
12. Pregnant or breastfeeding female or those with a positive pregnancy test or who will not use a medically acceptable contraceptive method from selection and during the study
13. Subject having used corticosteroid sporadically in the last 30 days whichever the route of administration, or any medication by ocular or nasal administration route
14. Subjects diagnosed with any ocular disease other than refractive error
15. Subject with history of ocular surgery, including laser refractive surgery
16. Subject using a contact lens within 7 days prior administration of the first dose
17. Intraocular pressure (IOP) ≥ 22 mmHg in either eye at screening or baseline
18. Presence of any corneal opacity or corneal fluorescein staining >0.5 grade using the modified Oxford scale in either eye at screening or baseline
19. Schirmer's test without anesthesia ≤ 9 mm/5 minutes in either eye at screening or baseline
20. Tear film break up time (TFBUT) < 8 seconds in either eye at screening or baseline Note: Alcoholic beverages should not be taken from 48 h before first drug administration until discharge from the Study center.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Director — Dompé SpA Milan
Locations (1):
- WCCT Global, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- rhNGF 20μg/mL: rhNGF 20μg/mL eye drop solution, formulation containing L-methionine as excipient.
  rhNGF 20μg/mL: Study Eye (For subjects randomized to rhNGF group) Day 1: One drop instilled into study eye (35 μL, corresponding to 0.70 μg of rhNGF).
  Day 2, 3, 4, 5, 6: One drop six times a day (every 2h) into study eye (210 μL, corresponding to 4.20 μg of rhNGF).
  Total dose in the study eye will be 31 drops (1085 μL, equivalent to 21.7 μg rhNGF) over 6 days.
Period: Overall Study
Arm/Group | rhNGF 20μg/mL | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 20μg/mL | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (10.82) | 33.1 (9.69) | 38.0 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs).
Description: TEAEs were defined as an adverse event (AE), which started after the first dose of study treatment. These comprise AEs during the treatment and follow-up period. For TEAE the number of events was provided.
Time Frame: On Day 1 (single dose scheme), Days 2-6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3), and Day 35-42 (FU 4)
Population: The safety population is represented by randomized subjects who received a dose of study medication in at least one eye. All 30 randomized subjects were included in the Safety population.
Measure: Number; unit: events
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
events | 27 | 9

2. Primary Outcome: Number of Treatment Emergent Adverse Events During First Dose Schedule (TEAEs Dose 1).
Description: TEAEs Dose 1 were defined as TEAEs, which started after the first dose of study treatment and before administration of the first dose at Treatment Day 2. For TEAE the number of events was provided.
Time Frame: During first dose schedule (TEAE Dose 1, which started after first dose of study treatment at Day 1 till before administration of the first dose at Treatment Day 2)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
events | 3 | 2

3. Primary Outcome: Number of Treatment Emergent Adverse Events During Second Dose Schedule (TEAEs Dose 2).
Description: TEAEs Dose 2 were defined as TEAEs, which started on/after the first dose at Treatment Day 2 and before Follow-Up Day 7 visit.
Time Frame: During second dose schedule (TEAE Dose 2, which started on/after the first dose at Treatment Day 2 till before Follow-Up Day 7 (FU1) visit
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
events | 16 | 4

4. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Ocular Tolerability Score in Study Eye: Single Dose
Description: Change from baseline in VAS ocular tolerability score in study eye at Treatment Day 2 predose (Tolerability of 1x0.70 μg rhNGF per day) for overall is presented. In this context, "Baseline" was defined as the pre-treatment assessment at the Baseline (D-1) visit.
  A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale.
Time Frame: at Treatment Day 2 pre-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale | 0.36 (1.325) | 0.24 (0.410)

5. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Ocular Tolerability Score in Study Eye: Multiple Dose
Description: Change from baseline in VAS ocular tolerability score in study eye at Day 2 8h, Day 3 predose, Day 6 pre-dose, Day 6 8h, Day 7 (FU1), Day 8 (FU2), Day 16 (FU3) (Tolerability of 6x0.70 μg rhNGF per day) for overall is presented. In this context, "Baseline" was defined as the pre-treatment assessment at the Baseline (D-1) visit.A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale.
Time Frame: at Day 2 8h, Day 3 predose, Day 6 pre-dose, Day 6 8h, Day 7 (FU1), Day 8 (FU2), Day 16 (FU3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Day 2 - 8h | 0.14 (0.882) | -0.09 (0.376)
  Day 3 - predose | 0.47 (0.673) | 0.14 (0.559)
  Day 6 - predose | 1.60 (5.091) | 0.17 (0.740)
  Day 6 - 8h | 1.85 (2.781) | -0.06 (0.358)
  FUI1 - 0h | 0.66 (3.828) | -0.13 (0.353)
  FUI2 - 8h | 0.40 (4.035) | -0.30 (0.474)
  FUI3 - 0h | -0.23 (1.470) | -0.01 (0.389)

6. Secondary Outcome: Number of Follow-Up AEs (FUAE)
Description: Follow-Up AEs (FUAE) were defined as TEAEs which start on or after Follow-Up Day 7 (FU1) visit
Time Frame: on or after Follow-Up Day 7 (FU1)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
events | 8 | 3

7. Secondary Outcome: Number of Ocular TEAEs by Eyes
Description: Ocular TEAEs were defined as an adverse event (AE) interesting the study or the non-study eye, which started after the first dose of study treatment. These comprise ocular AEs during the treatment and follow-up period. For these AE, the number of events was provided for the study eye and the non-study eye, separately.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
events
  study eye | 17 | 4
  non-study eye | 10 | 4

8. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP) by Eye Over All Visits
Description: IOP was performed using either Goldmann applanation tonometry after the instillation of a topical anaesthetic. IOP was measured in both eyes after completion of all other slit lamp examinations to avoid potential interference with the other evaluations.
Time Frame: on Day -1 and at Day 8 (Follow up [FU] 2) and Day 16 (FU3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
mmHg
  Study eye - FU 2 | -0.4 (2.70) | 0.5 (1.51)
  Study eye - FU 3 | -0.4 (3.03) | -0.3 (2.75)
  Non-study eye - FU 2 | -0.8 (1.92) | -0.3 (1.49)
  Non-study eye - FU 3 | -0.5 (2.48) | -0.5 (2.17)

9. Secondary Outcome: Change From Baseline in Visual Acuity Score for the Study Eye Over All Visits
Description: Values of Best-Corrected Distance Visual Acuity (BCDVA) scores were measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) score. The ETDRS charts use letters, or a geometric progression in letter size from line to line, under standardized lighting conditions. The patient starts at the top of the chart, or on the last row where he or she can read all of the letters, and reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified. Therefore, the higher the number of letters the higher the visual acuity. Changes in the ETDRS score from baseline are summarised for the study eye.
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
Letters
  Day 1 - 8h | 1.1 (3.03) | 0.6 (2.76)
  Day 2 - predose | 0.5 (3.47) | 0.4 (2.80)
  Day 2 - 8h | 1.8 (4.10) | 2.1 (2.77)
  Day 3 - predose | 0.8 (3.27) | 0.1 (3.87)
  Day 6 - predose | 1.6 (2.93) | 2.0 (3.43)
  Day 6 - 8h | 1.4 (3.72) | 2.5 (2.42)
  FU1 - 0h | 3.1 (3.62) | 2.4 (1.90)
  FU2 - 8h | 2.3 (3.06) | 1.5 (3.17)
  FU3 - 0h | 2.7 (3.59) | 1.4 (3.81)

10. Secondary Outcome: Change in Baseline in LogMAR [Derived as - Log (Snellen Equivalent Result)] for the Study Eye Over All Visits.
Description: LogMAR is the logarithm of the minimal angle of resolution. The LogMAR was derived as - log (Snellen Equivalent result). LogMAR values range from 1.6 (20/800 Snellen Equivalent) to -0.2 (20/12 Snellen Equivalent). The lower the LogMAR value, the better the visual acuity.
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
LogMAR
  Day 1 - 8 h | -0.025 (0.0547) | -0.019 (0.0757)
  Day 2 - predose | -0.015 (0.0785) | 0.010 (0.0536)
  Day 2 - 8h | -0.043 (0.0731) | -0.055 (0.0478)
  Day 3 - predose | -0.025 (0.0758) | -0.009 (0.0539)
  Day 6 - predose | -0.034 (0.0576) | -0.037 (0.0475)
  day 6 - 8h | -0.035 (0.0743) | -0.055 (0.0472)
  FU 1 - 0h | -0.073 (0.0820) | -0.055 (0.0478)
  FU2 - 8h | -0.049 (0.0684) | -0.018 (0.0594)
  FU3 - 0h | -0.054 (0.0751) | -0.028 (0.0901)

11. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) for the Study Eye Over All Visits..
Description: The TFBUT was performed after instillation of 5 μl of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner will monitor the integrity of the tear film, noting the time it takes to form lacunae (clear spaces in the tear film) from the time that the eye is opened after the last blink. The range of TFBUT normality in this trial is > 8' to 12' in either eye at screening or baseline.
  The longer the time the better the integrity of the tear film.
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
seconds
  Day 1 - 8h1 | -1.343 (2.0648) | -1.187 (1.5874)
  Day 2 - predose | -1.370 (1.9129) | -1.227 (1.3582)
  Day 2 - 8h | -1.000 (1.9806) | -1.761 (1.3983)
  Day 3 - predose | -0.612 (2.4824) | 0.344 (2.3712)
  Day 6 - predose | -0.593 (2.5198) | -1.442 (1.6595)
  Day 6 - 8h | -0.892 (2.0086) | -1.892 (1.5450)
  FU1 - 0h | -0.768 (2.0851) | 0.462 (1.3560)
  FU2 - 8h | -0.610 (1.8211) | -0.655 (2.4522)
  FU3 - 0h | -0.795 (2.1053) | -0.800 (1.4070)

12. Secondary Outcome: Change From Baseline in Overall National Eye Institute (NEI) Score for the Study Eye Over All Visits.
Description: Corneal Staining was derived as the sum of scores of the five corneal sectors (central, superior, inferior, nasal, and temporal) each of which was scored on a scale of 0-3, with a minimum score of 0 and a maximal score of 15 (sum > 3 out of 15 is abnormal).
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Day 1 - 8h1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 - predose | 0.5 (1.23) | 0.5 (1.27)
  Day 2 - 8h | 0.1 (0.22) | 0.0 (0.00)
  Day 3 - predose | 0.7 (1.79) | 0.6 (1.90)
  Day 6 - predose | 0.4 (1.35) | 0.0 (0.00)
  Day 6 - 8h | 0.0 (0.00) | 0.0 (0.00)
  FU1 - 0h | 0.7 (1.42) | 0.0 (0.00)
  FU2 - 8h | 0.1 (0.45) | 0.0 (0.00)
  FU3 - 0h | 0.1 (0.45) | 0.0 (0.00)

13. Secondary Outcome: Course of Visual Analogue Scale (VAS) Ocular Tolerability Score for the Study Eye Over All Visits.
Description: The course of VAS ocular tolerability score by eye over all visits was assessed. Only data "Overall" for study's eye are reported hereunder. A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale.
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Day 1 - 8h | 0.46 (0.890) | 0.09 (0.154)
  Day 2 - predose | 0.66 (1.739) | 0.31 (0.461)
  Day 2 - 8h | 0.81 (1.703) | 0.23 (0.358)
  Day 3 - predose | 1.14 (2.066) | 0.46 (0.499)
  Day 6 - predose | 2.26 (5.132) | 0.49 (0.661)
  Day 6 - 8h | 2.51 (7.089) | 0.26 (0.268)
  FU1 - 0h | 1.32 (3.548) | 0.19 (0.337)
  FU2 - 8h | 1.06 (3.727) | 0.01 (0.045)
  Fu3 - 0h | 0.44 (0.578) | 0.30 (0.428)

14. Secondary Outcome: Intraindividual Change in VAS Ocular Tolerability Scores Between Study Eye and Fellow (Non-study) Eye at All Study Visits
Description: Intraindividual differences between study eye and non-study (fellow) eye at all study visits were assessed. Data "overall" are reported hereunder.A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale.
Time Frame: On Day 1 (single dose scheme), Days 2,3,6 (multiple dose scheme), Day 7 (Follow-up [FU] 1), Day 8 (FU 2); Day 16 (FU 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Day 1 - 8h | 0.04 (0.258) | -0.06 (0.168)
  Day 2 - predose | 0.29 (1.024) | 0.10 (0.286)
  Day 2 - 8h | 0.11 (0.560) | -0.07 (0.205)
  Day 3 - predose | 0.54 (1.412) | 0.13 (0.519)
  Day 6 - predose | 1.16 (3.537) | 0.27 (0.698)
  Day 6 - 8h | 2.03 (6.942) | -0.09 (0.303)
  FU1 - 0h | 0.72 (2.823) | 0.04 (0.096)
  FU2 - 8h | 0.87 (3.697) | -0.03 (0.090)
  FU3 - 0h | 0.04 (0.346) | 0.00 (0.243)

15. Secondary Outcome: Kinetics of rhNGF Plasma Levels After Single-dose Administration and Multiple-dose Administration Through Enzyme-Linked Immunosorbent Assay I (ELISA I)
Description: Time points for rhNGF plasma levels measurement were the following:
  Day 1 (Pre-Dose, 0.5, 2, 4, 8, 9, 10, 11, 12, 14, 16 hr), Day 2 (Pre-Dose, 0.5, 2, 4, 6, 8, 10, 10.5, 11, 12, 13, 14, 16 hr), Day 3 (Pre-Dose, 2, 4, 6, 8, 10 hr), Day 4 Pre-Dose, Day 5 Pre-Dose, Day 6 (Pre-Dose, 4, 8, 10, 10.5, 11, 12, 13, 14, 16 hr), FU 1 0 hr, FU 2 (0 and 8 hr), and FU 3 0 hr.
  Values are reported for the single-dose regimen (Day 1) and the first day of the multiple-dose regimen (Day 2).
  From Day 1, most values were below the detectable level (i.e. <32 pg/ml). Values below this value are reported as not applicable (NA).
Time Frame: Day 1 (Pre-Dose, 0.5, 2, 4, 8, 9, 10, 11, 12, 14, 16 hr) and Day 2 (Pre-Dose, 0.5, 2, 4, 6, 8, 10, 10.5, 11, 12, 13, 14, 16 hr),
Population: PK-Set (PKS), defined as all subjects completing the PK sampling according to the study protocol and who did not show serious protocol deviations or non-compliance.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
pg/ml
  Day 1 - Pre-Dose | NA (94.16) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 0.5 hr | NA (83.06) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 2 hr | NA (66.73) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 4 hr | 35.69 (113.04) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 8 hr | NA (63.34) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 9 hr | NA (95.53) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 10 hr | 34.12 (94.85) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 11 hr | NA (82.12) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 12 hr | 33.10 (110.96) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 14 hr | NA (79.92) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 16 hr | 35.88 (117.91) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - Pre-Dose | 33.87 (113.95) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 0.5 hr | 32.30 (108.85) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 2 hr | NA (93.63) — values were below the detectable level (i.e. <32 pg/ml) | 1.02 (0)
  Day 2 - 4 hr | NA (77.01) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 6 hr | NA (83.02) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 8 hr | NA (90.77) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 10 hr | NA (90.40) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 10.5 hr | 34.68 (113.00) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 11 hr | 37.42 (120.37) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 12 hr | 32.22 (100.26) | NA (36.51) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 13 hr | NA (81.69) — values were below the detectable level (i.e. <32 pg/ml) | NA (34.96) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 14 hr | NA (96.51) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 16 hr | NA (101.13) — values were below the detectable level (i.e. <32 pg/ml) | NA (NA) — values were below the detectable level (i.e. <32 pg/ml)

16. Secondary Outcome: Kinetics of rhNGF Plasma Levels After Single-dose Administration and Multiple-dose Administration Through Enzyme-Linked Immunosorbent Assay II (ELISA II)
Description: Time points for rhNGF plasma levels measurement were the following:
  Day 1 (Pre-Dose, 0.5, 2, 4, 8, 9, 10, 11, 12, 14, 16 hr), Day 2 (Pre-Dose, 0.5, 2, 4, 6, 8, 10, 10.5, 11, 12, 13, 14, 16 hr), Day 3 (Pre-Dose, 2, 4, 6, 8, 10 hr), Day 4 Pre-Dose, Day 5 Pre-Dose, Day 6 (Pre-Dose, 4, 8, 10, 10.5, 11, 12, 13, 14, 16 hr), FU 1 0 hr, FU 2 (0 and 8 hr), and FU 3 0 hr.
  Values are reported for the single-dose regimen (Day 1) and the first day of the multiple-dose regimen (Day 2).
  From Day 1, most values were below the detectable level (i.e. <15 pg/ml). Values below this value are reported as not applicable (NA).
Time Frame: Day 1 (Pre-Dose, 0.5, 2, 4, 8, 9, 10, 11, 12, 14, 16 hr) and Day 2 (Pre-Dose, 0.5, 2, 4, 8, 9, 10, 10.5, 11, 12, 13, 14, 16 hr)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | rhNGF 20μg/mL | Placebo
Number analyzed (Participants) | 20 | 10
pg/ml
  Day 1 - Pre-Dose | 39.22 (105.51) | NA (36.08) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 0.5 hr | 36.28 (99.46) | NA (31.31) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 2 hr | 38.52 (105.06) | NA (28.70) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 4 hr | 39.43 (111.73) | NA (30.72) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 8 hr | 33.76 (90.93) | NA (31.69) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 9 hr | 35.27 (94.70) | NA (29.23) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 10 hr | 28.77 (68.13) | NA (23.69) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 11 hr | 34.87 (95.60) | NA (33.46) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 12 hr | 31.97 (86.13) | NA (32.38) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 14 hr | 34.23 (89.93) | NA (30.36) — values were below the detectable level (i.e. <32 pg/ml)
  Day 1 - 16 hr | 39.29 (111.35) | NA (25.93) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - Pre-Dose | 39.53 (113.26) | NA (32.57) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 0.5 hr | 34.35 (98.20) | NA (36.71) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 2 hr | 38.27 (103.68) | NA (37.84) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 4 hr | 35.51 (96.54) | 17.02 (41.93)
  Day 2 - 6 hr | 38.43 (106.00) | NA (31.75) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 8 hr | 33.90 (93.43) | NA (26.91) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 10 hr | 37.84 (102.03) | NA (27.13) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 10.5 hr | 39.64 (110.40) | NA (26.77) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 11 hr | 44.55 (121.82) | NA (26.51) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 12 hr | 37.81 (101.13) | NA (34.16) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 13 hr | 39.35 (104.93) | NA (33.78) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 14 hr | 37.31 (99.77) | NA (27.79) — values were below the detectable level (i.e. <32 pg/ml)
  Day 2 - 16 hr | 40.55 (118.50) | NA (16.32) — values were below the detectable level (i.e. <32 pg/ml)

ADVERSE EVENTS:
Time Frame: From Day -1 to Day 42
Arm/Group | rhNGF 20μg/mL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 10/20 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20μg/mL (N=20) | Placebo (N=10)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase incresed (Investigations) | 2 (2) | 1 (1)
Vital dye staining corneal present (Investigations) | 5 (9) | 3 (4)
Conjunctivitis (Infections and infestations) | 6 (6) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Catheter site oedema (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT03836859/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03836859/SAP_001.pdf